CLINICAL TRIAL: NCT02275052
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Effect of the Combination of Umeclidinium and Vilanterol on Exercise Endurance Time in Subjects With COPD
Brief Title: A Study to Evaluate the Effect of the Combination of Umeclidinium (UMEC) and Vilanterol (VI) on Exercise Endurance Time (EET) in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201317
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: shuttle walk test; umeclidinium; beta2-agonist; exercise endurance time; anticholinergic; combination product; vilanterol; exercise; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UMEC/VI 62.5/25mcg (Experimental): Participants will self-administer blinded UMEC/VI (62.5 mcg/25 mcg) each morning (once daily) as one inhalation from the double-blind DPI in one of the 2 treatment periods of 12 weeks. The treatment periods will be separated by a wash out period of 12-17 days.
  Interventions: Drug: UMEC/VI DPI; Drug: Albuterol/salbutamol MDI
- Placebo (Experimental): Participants will self-administer blinded placebo each morning (once daily) as one inhalation from the double-blind DPI in one of the 2 treatment periods of 12 weeks. The treatment periods will be separated by a wash out period of 12-17 days
  Interventions: Drug: Placebo DPI; Drug: Albuterol/salbutamol MDI

INTERVENTIONS:
Drug: UMEC/VI DPI — The DPI will contain a total of 30 doses. Each DPI will be comprised of two double-foil, laminate blister strips. Each blister of one strip will consist of 62.5mcg of UMEC blended with lactose and magnesium stearate while each blister of other strip will consist of 25 mcg of VI blended with lactose and magnesium stearate. Each actuation of the DPI will deliver the contents of one blister from each strip simultaneously
  Arms: UMEC/VI 62.5/25mcg
Drug: Placebo DPI — The placebo DPI, identical in appearance to the inhaler containing active study medication, will have two blister strips, each containing 30 blisters of lactose and magnesium stearate.
  Arms: Placebo
Drug: Albuterol/salbutamol MDI — Albuterol/salbutamol MDI (metered-dose inhaler) or nebules will be permitted throughout the study as rescue medication, for use as-needed. Albuterol/salbutamol will be sourced from local commercial stock or provided centrally from GlaxoSmithKline. Nebules will not be supplied.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, 2-period, complete block design cross-over study.

The purpose of this study is to evaluate the effect of UMEC/VI 62.5/25 microgram (mcg) on EET as measured by the Endurance Shuttle Walk Test (ESWT) compared to placebo. Additionally, the effect of UMEC/VI compared to placebo on lung function and lung volumes in COPD patients will be characterized.

Approximately 298 participants will be screened and, assuming 35% of these will not be eligible for randomization; approximately 194 participants will be randomized.

Eligible participants will be randomized 1:1 to one of 2 treatment sequences. In sequence 1 participants will receive UMEC/VI 62.5/25 mcg in Treatment Period 1 and placebo in Treatment Period 2. In sequence 2 participants will receive placebo in Treatment Period 1 and UMEC/VI 62.5/25 mcg in Treatment Period 2. Treatments will be delivered once-daily via a dry powder inhaler (DPI). Each treatment period will be for 12 weeks and will be separated by a wash out period of 12-17 days. The total duration of patient participation, including the Follow-Up will be approximately 30 weeks. All participants will be provided with albuterol for use on an "as needed (prn)" basis throughout the run-in, washout and study treatment periods while on investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Type of participant: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: 40 years of age or older at Visit 1.
* Gender: Male or female participants. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy. OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact): Abstinence; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Implants of levonorgestrel; Estrogenic vaginal ring; Percutaneous contraceptive patches; Intrauterine device (IUD) or intrauterine system (IUS) that meets the standard operating procedures (SOP); effectiveness criteria as stated in the product label; Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female participant's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the participant or review of the participant's medical history for study eligibility, as obtained via a verbal interview with the participant or from the participant's medical records; Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Diagnosis: A diagnosis of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years (number of pack years =[number of cigarettes per day /20] x number of years smoked [e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Severity of Disease: A pre- and post-albuterol Forced Expiratory Volume in One Second/Forced Vital Capacity (FEV1/FVC) ratio of <0.70 and a postalbuterol FEV1 of >=30% and <=70% of predicted normal values
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.
* Resting Lung Volumes: A resting FRC of >=120% of predicted normal FRC at Visit 1. Predicted values for FRC will be obtained using predicted normal values

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer in remission for <5 years are absolute exclusionary conditions. A participant who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Any participant who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any participant who has any condition besides COPD that is likely to affect respiratory function or the ability to perform exercise testing such as peripheral vascular disease should not be included in the study.
* Severe Hepatic Impairment: Patients with severe hepatic impairment (Child-Pugh class C) should be excluded unless, in the opinion of the investigator, the benefit is likely to outweigh the risk.
* Unstable or life threatening cardiac disease: Umeclidinium/vilanterol should be used with caution in participants with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV heart failure
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, sympathomimetic, lactose/milk protein or magnesium stearate.
* Antimuscarinic effects: Participants with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction should only be included if, in the opinion of the study physician, the benefit outweighs the risk.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1
* Lung Resection: Participants with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead Electrocardiogram (ECG): Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of participant eligibility. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the participant's medical history and exclude participants who would be at undue risk by participating in the trial. Participants with the following abnormalities are excluded from participation in the study: Atrial fibrillation with rapid ventricular rate >120 beats per minute (bpm); Sustained or nonsustained ventricular tachycardia; Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted)
* Medication Prior to Spirometry: Unable to withhold albuterol for the 4 hour period required prior to spirometry testing at each study visit
* Interactions: Concomitant administration with beta-blockers or strong Cytochrome P450 3A4 (CYP3A4) inhibitors is only permitted if, in the Investigator's opinion, the likely benefit outweighs the potential risk
* Medications prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids (12 weeks), systemic, oral or parenteral corticosteroids (Intra-articular and epidural corticosteroid injections are permitted) (6 weeks), antibiotics (for lower respiratory tract infection and/or COPD exacerbation) (6 weeks), long-acting beta agonist (LABA)/ inhaled corticosteroid (ICS) combination products if LABA/ICS therapy is discontinued completely (30 days), LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy (dose of ICS that is switched to must not exceed 1000mcg of fluticasone propionate or equivalent) (48 hours for the salmeterol or formoterol component 14 days for the vilanterol component), use of ICS at a dose >1000 microgram (mcg)/day of fluticasone propionate or equivalent (Use of ICS is permitted provided the dose does not exceed 1000mcg of fluticasone propionate or equivalent; ICS use not to be initiated or discontinued within 30 days prior to Visit 1 except for participants on LABA/ICS therapy who may discontinue LABA/ICS therapy as indicated and switch to ICS monotherapy) (30 days), initiation or discontinuation of ICS use (30 days), Phosphodiesterase 4 (PDE4) inhibitor (roflumilast) (14 days), Inhaled long acting beta2 agonists (LABA): salmeterol, formoterol (48 hours); olodaterol, indacaterol (14 days), Long-acting muscarinic antagonists (tiotropium, aclidinium, glycopyrronium, umeclidinium) (7 days), LAMA/LABA combination products (whichever mono component has the longest washout), theophyllines (48 hours), oral beta2-agonists (long-acting [48 hours], short-acting [12 hours]), inhaled short acting beta2-agonists (study provided prn albuterol/ is permitted during the study, except in the 4-hour period prior to spirometry testing) (4 hours), inhaled short-acting anticholinergics (permitted during the run-in period between Visits 1 and 4 and washout period between Visits 7 and 9. Participants must discontinue use of short-acting anticholinergics at least 4 hours before Visit 4 and Visit 9. Participants should not use short acting anticholinergics during the double-blind treatment periods) (4 hours), inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (4 hours), and any other investigational medication (30 days or within 5 drug half-lives [whichever is longer])
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol) via nebulized therapy
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Participants who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the Investigator, any participant who is unable to read and/or would not be able to complete a questionnaire
* Participation in Previous Exercise Studies: Participants who have previously been assigned a participant number (enrolled) in GlaxoSmithKline studies DB2114417 or DB2114418.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) who met the eligibility criteria at screening, entered the 11- to 25-day Run-in period followed by two 12-week Double-blind treatment periods that were separated by 12- to 17-day washout period. The total duration of participation, including the follow-up, was approximately 30 weeks.
Pre-assignment Details: A total of 374 par. were screened, of these, 10 par. were pre-screen failures, 132 par. were screen failures and 34 par. were run-in failures; 198 par. who were randomized into the study and received treatment were included in the Intent-to-Treat (ITT) Population.
Groups:
- Placebo Then UMEC/VI 62.5/25 µg: Participants received Placebo and then umeclidinium (UMEC)/ vilanterol trifenatate (VI) 62.5 micrograms (µg)/25 µg each morning (once daily) as one inhalation via the Dry Powder Inhaler (DPI) for 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed (prn)' basis throughout the run-in, washout and study treatment periods while on investigational product.
- UMEC/VI 62.5/25 µg Then Placebo: Participants received UMEC/ VI 62.5 µg/25 µg and then placebo each morning (once daily) as one inhalation via the DPI for 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed' basis throughout the run-in, washout and study treatment periods while on investigational product.
- Period 2: UMEC/VI 62.5/25 µg Then Placebo: Participants received UMEC/VI 62.5 µg/25 µg and then Placebo each morning (once daily) as one inhalation via the Dry Powder Inhaler (DPI) for 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed (prn)' basis throughout the run-in, washout and study treatment periods while on investigational product.
- Period 2: Placebo Then UMEC/VI 62.5/25 µg: Participants received placebo and then UMEC/VI 62.5 µg/25 µg each morning (once daily) as one inhalation via the DPI for 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed' basis throughout the run-in, washout and study treatment periods while on investigational product.
Period: Period 1: Treatment Period 1 (12 Weeks)
Arm/Group | Placebo Then UMEC/VI 62.5/25 µg | UMEC/VI 62.5/25 µg Then Placebo | Period 2: UMEC/VI 62.5/25 µg Then Placebo | Period 2: Placebo Then UMEC/VI 62.5/25 µg
Started | 99 | 99 | 0 | 0
Completed | 90 | 93 | 0 | 0
Not Completed | 9 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Met protocol-defined stopping criteria | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Period: Washout Period (12-17 Days)
Arm/Group | Placebo Then UMEC/VI 62.5/25 µg | UMEC/VI 62.5/25 µg Then Placebo | Period 2: UMEC/VI 62.5/25 µg Then Placebo | Period 2: Placebo Then UMEC/VI 62.5/25 µg
Started | 90 | 93 | 0 | 0
Completed | 86 | 93 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Period: Period 2: Treatment Period 2 (12 Weeks)
Arm/Group | Placebo Then UMEC/VI 62.5/25 µg | UMEC/VI 62.5/25 µg Then Placebo | Period 2: UMEC/VI 62.5/25 µg Then Placebo | Period 2: Placebo Then UMEC/VI 62.5/25 µg
Started | 0 | 0 | 93 | 86
Completed | 0 | 0 | 88 | 72
Not Completed | 0 | 0 | 5 | 14
Not completed — Adverse Event | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 6
Not completed — Met Protocol-defined Stopping Criteria | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- UMEC/VI 62.5/25 mcg and Placebo in One of the Two Sequences: Par. received a sequence consisting of the following 2 treatments: One inhalation of UMEC/VI 62.5/25 mcg or placebo once daily using a DPI. Each treatment was self-administered in the morning for 12 weeks. The treatments were separated by a 12 to 17 day washout period; all par. were provided with albuterol for use on an 'as needed' basis throughout the run-in, washout and study treatment periods while on investigational product.
Arm/Group | UMEC/VI 62.5/25 mcg and Placebo in One of the Two Sequences
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 104
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 19
  White-White/Caucasian/European Heritage | 179

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Exercise Endurance Time (EET) Post-dose at Week 12 of Each Treatment Period
Description: EET post-dose at W12 is defined as the EET obtained 3 hours after dosing at W12. EET was measured using the externally paced field walking test called endurance shuttle walk test (ESWT). Change from BL in EET at W12 was analyzed using a repeated measures model with covariates of period walking speed, mean walking speed, period, trt, visit (Day 2, W6 and W12), smoking status, visit by period walking speed, visit by mean walking speed and visit by trt interactions. BL was the EET assessment obtained prior to dosing on Day 1 of each period. The mean walking speed for each par. is the mean of the levels used for the ESWT in each of the two trt periods. Period walking speed for each par. and trt period is the difference between the level for that par. and period and the mean walking speed for that par. Intent-to-treat (ITT) Population: all randomized par., excluding those who were randomized in error, and par. who discontinued trt (off-trt).
Time Frame: Baseline (BL) and at Week (W) 12 of each treatment (trt) period (up to Week 30)
Population: ITT Population including off-treatment data. Number of par. represent those with data available at the time point; however, all par. in the ITT population without missing covariate information and with at least one post Baseline measurement are included.
Measure: Least Squares Mean (Standard Error); unit: Seconds (s)
Groups:
- UMEC/VI 62.5/25 mcg: Participants received umeclidinium (UMEC)/ vilanterol trifenatate (VI) 62.5 mcg/25 mcg each morning (once daily) as one inhalation via the DPI in one of the 2 treatment periods of 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed (prn)' basis throughout the run-in, washout and study treatment periods while on investigational product.
- Placebo: Participants received placebo each morning (once daily) as one inhalation via the DPI in one of the 2 treatment periods of 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed' basis throughout the run-in, washout and study treatment periods while on investigational product.
Arm/Group | UMEC/VI 62.5/25 mcg | Placebo
Number analyzed (Participants) | 172 | 157
Seconds (s) | -2.06 (9.286) | -5.37 (9.680)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg vs Placebo; Test type: Superiority or Other; p = 0.790, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 3.31, 95% CI 2-sided [-21.12 to 27.74] — Least squares mean change difference=UMEC/VI 62.5/25 µg minus Placebo

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 12 of Each Treatment Period
Description: Trough FEV1 is a measure of lung function and is defined as the mean of FEV1 values obtained 23 and 24 hours after dosing on the previous day. Trough FEV1 measurements were taken electronically by spirometry on Day 2, Week 6 and Week 12. Baseline was the assessment recorded before dosing on Day 1 of each period. Mean Baseline is the mean of the Baselines for each participant. Period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Analysis was performed using a repeated measures model and the following covariates were included: period Baseline, mean Baseline, period, treatment, visit, smoking status, visit by period Baseline, visit by mean Baseline and visit by treatment interactions.
Time Frame: Baseline and at Week 12 of each treatment period (up to Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg | Placebo
Number analyzed (Participants) | 175 | 164
Liters | 0.173 (0.0152) | -0.034 (0.0156)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.206, 95% CI 2-sided [0.167 to 0.246] — Least squares mean change difference=UMEC/VI 62.5/25 µg minus Placebo

3. Secondary Outcome: Change From Baseline in Functional Residual Capacity (FRC) 3 Hours Post-dose at Week 12 of Each Treatment Period
Description: FRC is defined as the amount of air still left in the lungs after breathing out normally. Standard body plethysmography techniques were used for lung volumes. Baseline is the assessment recorded before dosing on Day 1 of each period. Mean Baseline is the mean of the Baselines for each participant. Period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. FRC 3 hours post-dose was measured from the value obtained 3 hours after dosing on Day 2 and Week 12. Analysis was performed using a repeated measures model and the following covariates were included: period Baseline, mean Baseline, period, treatment, visit, smoking status, visit by period Baseline, visit by mean Baseline and visit by treatment interactions.
Time Frame: Baseline and at Week 12 of each treatment period (up to Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg | Placebo
Number analyzed (Participants) | 178 | 162
Liters | -0.457 (0.0531) | -0.111 (0.0557)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = -0.346, 95% CI 2-sided [-0.487 to -0.204] — Least squares mean change difference=UMEC/VI 62.5/25 µg minus Placebo

4. Secondary Outcome: Change From Baseline in Inspiratory Capacity (IC) 3 Hours Post-dose at Week 12 of Each Treatment Period
Description: IC is defined as the maximum amount of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Standard body plethysmography techniques were used for lung volumes. Baseline is the IC value recorded pre-dose on Day 1 of each treatment period. Mean Baseline is the mean of the Baselines for each par. Period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each par. IC 3-hours post-dose was measured from the value obtained 3 hours after dosing on Day 2 and Week 12. Analysis performed using a repeated measures model with covariates of period Baseline, mean Baseline, period, treatment, visit (Day 2 or Week 12), smoking status, visit by period Baseline, visit by mean Baseline and visit by treatment interactions.
Time Frame: Baseline and at Week 12 of each treatment period (up to Week 30)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 mcg | Placebo
Number analyzed (Participants) | 178 | 162
Liters | 0.225 (0.0266) | -0.034 (0.0278)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 mcg vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.259, 95% CI 2-sided [0.194 to 0.324] — Least squares mean change difference=UMEC/VI 62.5/25 µg minus Placebo

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of investigational product and until one day after last dose (approximately Week 25).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population.
Groups:
- UMEC/VI 62.5/25 mcg: Participants received umeclidinium (UMEC)/ vilanterol trifenatate (VI) 62.5 mcg/25 mcg each morning (once daily) as one inhalation via the Dry Powder Inhaler (DPI) in one of the 2 treatment periods of 12 weeks. The treatment periods were separated by a washout period of 12-17 days; all par. were provided with albuterol for use on an 'as needed (prn)' basis throughout the run-in, washout and study treatment periods while on investigational product.
Arm/Group | UMEC/VI 62.5/25 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/198 | 4/198
Other Adverse Events (participants affected / at risk) | 0/198 | 0/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 mcg (N=198) | Placebo (N=198)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.